CLINICAL TRIAL: NCT06469762
Title: The Short-Term Effects of Dry Cupping the Lumbar Paraspinal Muscles in Individuals With Non-specific Low Back Pain: A Single-Blind Randomized Trial
Brief Title: The Short-Term Effects of Dry Cupping the Lumbar Paraspinal Muscles in Individuals With Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LakeheadU-Scavarelli
Record Dates: First submitted 2024-05-03; First posted 2024-06-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Non-specific Low Back Pain
Keywords: Dry Cupping

STUDY DESIGN:
Intervention Model Description: Randomized trial with an intervention and placebo group. 2 x 2 x 3 mixed design, measures will be taken pre- and post-treatment in all 3 treatment sessions.
Who Masked: Participant
Masking Description: Participants will be unaware of their treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Individuals in this condition will receive treatment using plastic cups with two 2 mm holes drilled in either side of them, for all three treatment sessions.
  Interventions: Other: Placebo Dry Cupping
- Intervention (Experimental): Individuals in this condition will receive treatment using regular plastic cups, for all three treatment sessions.
  Interventions: Other: Dry Cupping

INTERVENTIONS:
Other: Dry Cupping — Dry cupping treatment session, using 4 regular plastic cups on the lumbar spine for 10 minutes.
  Arms: Intervention
Other: Placebo Dry Cupping — Dry cupping treatment session, using 4 plastic cups with two 2 mm holes drilled in either side of them, on the lumbar spine for 10 minutes.
  Arms: Placebo

SUMMARY:
This pilot study will investigate the effects of dry cupping the lumbar paraspinal muscles on lumbar spine on range of motion (ROM), blood flow as indicated by skin temperature, subjective pain, pressure pain threshold, perceived treatment effect and overall function in individuals experiencing Non-specific low back pain (NSLBP). The intervention will occur across three treatment sessions, scheduled approximately 48 hours apart. Both an intervention and placebo group will be used an a pre-/post- comparison will be conducted.

DETAILED DESCRIPTION:
Once the ethics approval has been provisionally granted, the pilot study will be registered as a randomized clinical trial with finalized and approved protocol. After the registration has been completed, prospective participant recruitment will begin. The study recruitment will occur through the use of recruitment posters around Lakehead University and posted on the investigator's Instagram© and Facebook© pages. In addition, local chiropractic and physiotherapy clinics will be contacted to inquire about recruiting within their clinics and through their social media platforms. The investigators are targeting at least 60 participants to be recruited who are experiencing NSLBP, are otherwise healthy, are within 18-55 years of age, and consent to be a participant. Should the participant be currently receiving treatment for NSLBP or another musculoskeletal condition, a wash out period of 2 days (48 hours) will be ensured between their treatment and study participation. Exclusion criteria will include any individual with a previous or scheduled surgery to the lower body which may affect their hip and/or knee ROM, previously experienced trauma to the low back area, are diagnosed with a specific low back or lower body condition (i.e., spondylolisthesis, spinal stenosis, osteoporosis, or intervertebral disk derangement), are diagnosed with cancer, are experiencing referred leg symptoms, are confirmed or suspected to be pregnant, or with a confirmed or suspected blood/blood clotting disorder (i.e., hemophiliac).

After potential participants contact the investigator regarding their interest in the pilot study, a detailed information letter will be provided to them. The information letter will include details pertaining to the pilot study including the purpose, procedures, duration, potential session availabilities, and the location at which the research will take place. If the prospective participant is still interested in engaging in the pilot study, they will arrange an appropriate time to meet with the investigator for data collection. Three sessions will be scheduled, each approximately 48 hours apart (e.g., Monday, Wednesday and Friday). Each session will last about 60 minutes and will take place at Lakehead University in the School of Kinesiology Sanders Building in room SB-1025.

Participants will be randomly assigned to either a placebo or intervention group, which will be decided prior to the first session. Should the participant be in the placebo group and wish to receive treatment, they will be offered this opportunity upon the completion of the data collection session. In the first session, the potential participant will review and sign the provided consent form. The investigator will also explain the ability to withdraw from the pilot study at any time without penalty. After informed consent has been given, the participant will then complete the Get Active Questionnaire (GAQ) and a Participant Demographic form which will include information related to their gender, sex, age, height, and body mass. Should the participant respond "Yes" to any question on the GAQ, they must be cleared by their medical provider prior to participation.

At this point the intervention will begin, the participant will be asked to lay prone on the examination table, with their lumbar spine exposed. The investigator will landmark the L1 and L5 vertebrae and mark this location with a washable, skin safe marker. This will be located by palpating for the iliac crests and following them directly inward to landmark the spinous processes of L4. From there, L5 will be marked one thumb-width downward from the spinous process of L4, and L1 will be marked three thumb-widths up the spine after palpating the spinous processes of the respective vertebral bodies. From there, the investigator will measure 3 centimeters (cm) on each side of the landmarked spinous processes of L1 and L5, using the measuring tape. This will be done to standardize the location of the inclinometers, and all four locations will be marked using a marker. Next, the participant will be asked to identify their primary location of LBP (by pointing to the area; e.g., right side of L3), this area will be marked using a marker and will represent problem area one (P1). The participant will then be asked to name their secondary location of LBP (by pointing to the area; e.g., left side of L4), this area will be marked using a marker and will represent problem area two (P2). After the locations have been marked, baseline measurements will be taken. The skin temperature of the lumbar spine will be taken using the Maximum™ Laser Thermometer at P1 and P2 and the mean skin temperature will be calculated and recorded to the nearest tenth of a degree. Following that, the pressure pain threshold will be measured using the Wagner Force One™ Digital Force Gauge. Firstly, the participant will be asked to identify an area of no pain (e.g., the deltoid, triceps, or gastrocnemius), the pressure pain threshold will be measured at the indicated location, and the result will be recorded. This will be done by applying the tip of the Wagner Force One™ Digital Force Gauge perpendicular to the indicated area and applying a gradually increasing amount of pressure. The participant will be asked to indicate when the pressure sensation on the area transitions to a sensation of pain. At this point, the value indicated on the algometer will be recorded and the pressure will be removed. This will be used to establish a baseline in an area of no pain, and to familiarize the participant with the measurement tool. Next, measurements will be taken at P1 and P2, and the two measurements will be recorded to the nearest tenth of a Newton (N). Next, the participant will be asked to stand, and two inclinometers will be placed on the L1 and L5 landmarks on the ride side of the spine. The participant will be instructed to bend forward as far as comfortably possible. The mean of the two values measured by the inclinometers will be recorded to the nearest tenth of a degree. This will be completed again with the inclinometers on the left side and the mean of both the L1 and L5 values will be recorded. Following the measurements on both sides, the average of the right and left side measurements will be recorded. Finally, the participant will complete the Sit and Reach Test using the Sit and Reach Device. The Sit and Reach Test will be conducted by instructing the participant to remove their shoes and sitting on the floor with their back against a wall and legs out straight in long sitting. The feet will be placed into the foot pedals and their hands will be clasped together and resting on the metal measuring piece. The participant will be asked to keep their legs flat, and feet pressed against the pedals. They will then be asked to reach forward as far as possible, pushing the metal measuring piece with their fingertips. After 3 warm-up tries, the participant will hold the fourth trial for 3 seconds and the measurement will be recorded to the nearest tenth of a cm. The participant will also complete the Numeric Pain Rating Scale (NPRS) and be asked to indicate their current low back pain on a scale from 0 (no pain) to 10 (worst possible pain). Finally, the participant will complete the Roland-Morris Questionnaire, to assess their overall function. The questionnaire will be scored by the investigator and the result will be recorded. Further information regarding psychometric properties of this tool will be provided in the Outcome Measures section.

Following the baseline measurements, the cupping treatment will begin. Once again, the participant will be asked to lay prone on the examination table. The investigator will apply a light layer of skin adhesive spray to the participant's lumbar spine at the 4 cupping locations. This will be used to improve suction. Four medium sized Hansol© plastic cups will be placed superior and inferior to P1 and P2 (i.e., superior to P1, inferior to P1, superior to P2, and inferior to P2). Those in the placebo group will receive cups with holes punctured in them, so that the suction is immediately released, while the adhesive spray will ensure the cups remain in place and do not change the sensation for the participant. Each cup will be pumped three times using the hand pump for consistent suction (465 mmHg of pressure). The cups will be left in a static position for a total of 10 minutes. After the treatment is concluded, the suction will be released, and the cups will be removed and placed into a bin to be later disinfected by the hydrogen peroxide solution as per the manufacturer's instructions.

Immediately following the cupping intervention, the skin temperature of P1 and P2 will be taken again using the Maximum™ (Model N08064) Laser Thermometer and the mean will be recorded. The pressure pain threshold will once again be measured using the Wagner Force One™ Digital Force Gauge at P1 and P2 as well as the non-painful site, and the dual inclinometry lumbar flexion and Sit and Reach Test will also be repeated, and the post intervention results will be recorded as described previously. The participant will also complete the NPRS once again and be asked to rate their current low back pain on a scale from 0 to 10. Next, they will complete the Roland-Morris Questionnaire, to assess their overall function, and finally, they will complete the Patient Global Impression of Change Scale (PGICS) and be asked to reflect on their treatment experience and indicate if their condition is "very much improved" (1) to "very much worse" (7). Further information regarding psychometric properties of this tool will be provided in the Outcome Measures section.

The participant will be thanked for their involvement and offered to receive a copy of the results at the completion of the pilot study. If the participant wishes, their email will be recorded to forward the results at a later date. Once the participant has left, the investigator will disinfect the table, inclinometer, and Sit and Reach Device using a disinfectant spray. The cups will be washed in a bin of warm water with dish detergent. After they are rinsed, they will be dried with paper towel, and taken and placed into the pre-mixed 3% hydrogen peroxide solution for 10 minutes as per the manufacturer's instructions. The solution will be made by combining one part 35% hydrogen peroxide with 11 parts water. After 10 minutes, the cups will be removed and set aside to dry before being used on the next participant.

The procedures will remain the same for both the individuals in the intervention and placebo condition, however, those in the placebo condition will receive cups with two 2 millimeter (mm) holes drilled in either side of them, so that the suction is immediately released upon application.

In the second and third sessions, the procedures will be repeated as previously described, with the exclusion of the consent form, GAQ, and Patient Demographic Form.

ELIGIBILITY:
Inclusion Criteria:

* Males and females;
* Between the ages of 18 - 55 years;
* Experiencing NSLBP; and
* Otherwise healthy, and successful completion of the GAQ (Should the participant be currently receiving treatment for NSLBP for another musculoskeletal condition, a wash out period of 2 days (48 hours) will be ensured between their treatment and study participation).

Exclusion Criteria:

* Any individual with a specific low back or lower body condition (e.g., i.e., spondylolisthesis, spinal stenosis, osteoporosis, intervertebral disk derangement);
* Any individual with a previous or scheduled surgery to the lower body, which may affect their hip and/or knee ROM;
* Any individual with previous trauma to the lower back area;
* Any individual who is diagnosed with cancer;
* Any individual experiencing referred leg symptoms;
* Any individual who is confirmed or suspected to be pregnant; and
* Any individual with a confirmed or suspected blood/blood clotting disorder (i.e., hemophiliac).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale (NPRS) | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  A self-administered pain questionnaire that requires individuals to reflect on their current level of pain on a scale from 0 (no pain) to 10 (the worst possible pain). This is one of the most common methods of assessing patient subjective pain perception as it is easily understood and simple to interpret. This tool has demonstrated excellent reliability (r=.99) for assessing musculoskeletal pain and a very high intraclass correlation coefficient (ICC=.95). The minimal detectable change (MDC) for this tool is 1.33 points. This score indicates the minimal change in NPRS score needed to assume a true change.
Algometry | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  A Wagner Force One™ Digital Force Gage will be used to measure the pressure pain threshold. It is considered the gold standard for measuring subjective pain. The pressure pain threshold will first be measured in a non-painful area identified by the participant (e.g. deltoid) to establish a baseline, which will be recorded. Next, it will be measured at P1 and P2 and the two measurements will be taken and recorded, both pre- and post-intervention. This tool has demonstrated good to excellent intra-rater (r=.75-.99) and good to excellent interrater (r=.81-.99) reliability in measuring low back pain. The MDC for this tool is 47.2 kilopascals (kPa).

SECONDARY OUTCOMES:
The Sit and Reach Test | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  A method for assessing lumbar spine ROM and will be used to make comparisons between pre- and post-intervention. This test requires the participant to sit on the floor with their feet pressed against the pedals on the Sit and Reach Device. They must then reach forward as far as possible while pushing a metal measuring piece with their fingertips. This tool has demonstrated a moderate interclass correlation coefficient (r=.57-.74) and an excellent intraclass correlation coefficient (r=.92), indicating its high reliability. The MDC for the Sit and Reach Test is between 1.13 cm and 1.74 cm. This value indicates the minimal change in the Sit and Reach score needed to assume a true change.
Lumbar flexion inclinometry | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  A method of measuring lumbar spine flexion ROM. The use of dual inclinometers allows for one to be placed at both L1 and L5 and an average measurement to be taken. For this measure, the participant will be required to bend forward as far as comfortably possible, and the mean value will be recorded. This will be completed for both the right and left sides at the locations of the cups. This tool has demonstrated excellent interrater (r=.88-.94), excellent intra-rater (r=.90-.91) and excellent test-retest (r=.91-.93) reliability for measuring thoracolumbar spine ROM in individuals with LBP. The MDC for inclinometry is between 1.50° and 3.41°. This score indicates the minimal change in the inclinometry value needed to assume a true change.
Skin Temperature | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  The Maximum™ (Model N08064) Laser Thermometer will be used to measure lumbar spine skin temperature pre- and post-treatment. This will be measured in degrees Celsius (ºC) before and immediately after the cupping treatment at P1 and P2. The mean of the measurements will be taken and recorded.
The Patient Global Impression of Change Scale (PGICS) | Immediately after intervention #1, immediately after intervention #2, immediately after intervention #3
  A self-report questionnaire that requires individuals to reflect on their overall perception of a treatment or intervention. It allows individuals to make a comparison between their condition pre- and post-intervention and rate it from 1 (very much improved) to 7 (very much worse). It is a standardized method of measure patient report outcomes with a high test-retest reliability (ICC=.84) in patients with LBP.
Roland-Morris Questionnaire | Pre-intervention #1, immediately after intervention #1, pre-intervention #2, immediately after intervention #2, pre-intervention #3, immediately after intervention #3
  A validated measure commonly used by practitioners to assess physical disability caused by low back pain. It is a self-report questionnaire that is scored to obtain a functional score. The patient is asked to indicate when a statement applies to that specific day, this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 24 (max. disability). This tool has demonstrated excellent intra-rater reliability (ICC=.91), with moderate internal (r=.71) and external (r=.54) responsiveness. The MDC for this tool is 5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Almeida Silva HJ, Avila MA, Castro KMS, Pinheiro YT, Lins CAA, Medeiros Barbosa G, de Souza MC. Exploring patient experiences of participating in a real and sham dry cupping intervention for nonspecific low back pain: A qualitative study. PLoS One. 2022 May 19;17(5):e0268656. doi: 10.1371/journal.pone.0268656. eCollection 2022. PMID 35587506
- [Background] Al-Qahtani SG, Alsulami BA. Prevalence and predictors of use of cupping among patients attending a primary care center in Riyadh, Saudi Arabia. J Family Med Prim Care. 2023 Feb;12(2):376-382. doi: 10.4103/jfmpc.jfmpc_1615_22. Epub 2023 Feb 28. PMID 37090992
- [Background] Amundsen PA, Evans DW, Rajendran D, Bright P, Bjorkli T, Eldridge S, Buchbinder R, Underwood M, Froud R. Inclusion and exclusion criteria used in non-specific low back pain trials: a review of randomised controlled trials published between 2006 and 2012. BMC Musculoskelet Disord. 2018 Apr 12;19(1):113. doi: 10.1186/s12891-018-2034-6. PMID 29650015
- [Background] Ayala F, Sainz de Baranda P, De Ste Croix M, Santonja F. Reproducibility and criterion-related validity of the sit and reach test and toe touch test for estimating hamstring flexibility in recreationally active young adults. Phys Ther Sport. 2012 Nov;13(4):219-26. doi: 10.1016/j.ptsp.2011.11.001. Epub 2012 Jan 23. PMID 23068896
- [Background] Bobos P, Ziebart C, Furtado R, Lu Z, MacDermid JC. Psychometric properties of the global rating of change scales in patients with low back pain, upper and lower extremity disorders. A systematic review with meta-analysis. J Orthop. 2020 Feb 10;21:40-48. doi: 10.1016/j.jor.2020.01.047. eCollection 2020 Sep-Oct. PMID 32082038
- [Background] Boyd BS. Measurement properties of a hand-held inclinometer during straight leg raise neurodynamic testing. Physiotherapy. 2012 Jun;98(2):174-9. doi: 10.1016/j.physio.2011.04.352. Epub 2011 Jun 8. PMID 22507369
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Dimitriadis Z, Parintas I, Karamitanis G, Abdelmesseh K, Koumantakis GA, Kastrinis A. Reliability and Validity of the Double Inclinometer Method for Assessing Thoracolumbar Joint Position Sense and Range of Movement in Patients with a Recent History of Low Back Pain. Healthcare (Basel). 2022 Dec 29;11(1):105. doi: 10.3390/healthcare11010105. PMID 36611565
- [Background] Duniec L, Nowakowski P, Kosson D, Lazowski T. Anatomical landmarks based assessment of intravertebral space level for lumbar puncture is misleading in more than 30%. Anaesthesiol Intensive Ther. 2013 Jan-Mar;45(1):1-6. doi: 10.5603/AIT.2013.0001. PMID 23572300
- [Background] Fang H, Ho IMK. Intraday reliability, sensitivity, and minimum detectable change of national physical fitness measurement for preschool children in China. PLoS One. 2020 Nov 20;15(11):e0242369. doi: 10.1371/journal.pone.0242369. eCollection 2020. PMID 33216780
- [Background] Gallasch CH, Alexandre NM. The measurement of musculoskeletal pain intensity: a comparison of four methods. Rev Gaucha Enferm. 2007 Jun;28(2):260-5. PMID 17907648
- [Background] Lemmink KA, Kemper HC, de Greef MH, Rispens P, Stevens M. The validity of the sit-and-reach test and the modified sit-and-reach test in middle-aged to older men and women. Res Q Exerc Sport. 2003 Sep;74(3):331-6. doi: 10.1080/02701367.2003.10609099. No abstract available. PMID 14510299
- [Background] Markowski A, Sanford S, Pikowski J, Fauvell D, Cimino D, Caplan S. A pilot study analyzing the effects of Chinese cupping as an adjunct treatment for patients with subacute low back pain on relieving pain, improving range of motion, and improving function. J Altern Complement Med. 2014 Feb;20(2):113-7. doi: 10.1089/acm.2012.0769. Epub 2013 Dec 3. PMID 24299469
- [Background] Mayorga-Vega D, Merino-Marban R, Viciana J. Criterion-Related Validity of Sit-and-Reach Tests for Estimating Hamstring and Lumbar Extensibility: a Meta-Analysis. J Sports Sci Med. 2014 Jan 20;13(1):1-14. eCollection 2014 Jan. PMID 24570599
- [Background] Nussbaumer S, Leunig M, Glatthorn JF, Stauffacher S, Gerber H, Maffiuletti NA. Validity and test-retest reliability of manual goniometers for measuring passive hip range of motion in femoroacetabular impingement patients. BMC Musculoskelet Disord. 2010 Aug 31;11:194. doi: 10.1186/1471-2474-11-194. PMID 20807405
- [Background] Salemi MM, Gomes VMDSA, Bezerra LMR, Melo TMS, Alencar GG, Montenegro IHPM, Calado APM, Montenegro EJN, Siqueira GR. Effect of Dry Cupping Therapy on Pain and Functional Disability in Persistent Non-Specific Low Back Pain: A Randomized Controlled Clinical Trial. J Acupunct Meridian Stud. 2021 Dec 31;14(6):219-230. doi: 10.51507/j.jams.2021.14.6.219. PMID 35770601
- [Background] Stephens SL, DeJong Lempke AF, Hertel J, Saliba S. Clinical usage, application procedures, and perceived effectiveness of cupping therapy among healthcare professionals in the United States: A cross-sectional survey. Complement Ther Clin Pract. 2022 Aug;48:101610. doi: 10.1016/j.ctcp.2022.101610. Epub 2022 Jun 3. PMID 35717744
- [Background] Volpicelli Leonard K, Robertson C, Bhowmick A, Herbert LB. Perceived Treatment Satisfaction and Effectiveness Facilitators Among Patients With Chronic Health Conditions: A Self-Reported Survey. Interact J Med Res. 2020 Mar 6;9(1):e13029. doi: 10.2196/13029. PMID 32141836
- [Background] Wang YT, Qi Y, Tang FY, Li FM, Li QH, Xu CP, Xie GP, Sun HT. The effect of cupping therapy for low back pain: A meta-analysis based on existing randomized controlled trials. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1187-1195. doi: 10.3233/BMR-169736. PMID 28946531
- [Background] Wood S, Fryer G, Tan LLF, Cleary C. Dry cupping for musculoskeletal pain and range of motion: A systematic review and meta-analysis. J Bodyw Mov Ther. 2020 Oct;24(4):503-518. doi: 10.1016/j.jbmt.2020.06.024. Epub 2020 Jul 30. PMID 33218554
- [Background] Bhattacharyya A, Hopkinson LD, Nolet PS, Srbely J. The reliability of pressure pain threshold in individuals with low back or neck pain: a systematic review. Br J Pain. 2023 Dec;17(6):579-591. doi: 10.1177/20494637231196647. Epub 2023 Aug 26. PMID 37969131
- [Background] Salom-Moreno J, Ortega-Santiago R, Cleland JA, Palacios-Cena M, Truyols-Dominguez S, Fernandez-de-las-Penas C. Immediate changes in neck pain intensity and widespread pressure pain sensitivity in patients with bilateral chronic mechanical neck pain: a randomized controlled trial of thoracic thrust manipulation vs non-thrust mobilization. J Manipulative Physiol Ther. 2014 Jun;37(5):312-9. doi: 10.1016/j.jmpt.2014.03.003. Epub 2014 May 28. PMID 24880778